CLINICAL TRIAL: NCT01266564
Title: A Non-interventional Multicenter Study of First-line Avastin® (Bevacizumab) in Combination With Chemotherapy in Patients With Metastatic Colorectal Cancer
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25198
Record Dates: First submitted 2010-12-20; First posted 2010-12-24 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will assess the progression-free survival, overall response and safety of Avastin (bevacizumab) in combination with chemotherapy in a real life setting in patients with metastatic colorectal cancer. Data will be collected from patients for approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age >/=18 years
* Proven metastatic colorectal carcinoma
* Patients have measurable disease
* Patients are eligible to receive first-line Avastin
* Patients have signed data release form

Exclusion Criteria:

* Contra-indication to receive Avastin according to the local labeling
* Participation in a clinical study within 30 days prior to enrolment
* Patients have any other primary cancer
* Concomitant treatment with other biologics
* History of other malignant disease in the past 5 years except basal cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients receiving Avastin in combination with chemotherapy
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2010-09-03 (Actual); Primary Completion 2015-07-10 (Actual); Study Completion 2015-07-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival in a real life setting assessed by computer tomography | Approximately 2 years

SECONDARY OUTCOMES:
Overall response rate assessed by computer tomography | Approximately 2 years
Response of Avastin according to the sites of metastases assessed by computer tomography | Approximately 2 years
Chemotherapy regimens used in combination with Avastin | Approximately 2 years
Patient demographics eligible to receive Avastin | Approximately 2 years
Safety: incidence of adverse events | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Lebanon (14):
  - American University of Beirut - Medical Center, Beirut
  - Saint George Hospital; Haematology-Oncology, Beirut
  - Hotel Dieu de France; Oncology, Beirut
  - Mount Lebanon Hospital, Beirut
  - Beirut Governmental University Hospital, Beirut
  - Al-Rassoul Al-Aazam Hospital, Beirut
  - Lebanese Hospital Geitaoui, Beirut
  - Middle East Inst. of Health; Oncology, Beirut
  - Notre Dame Des Secours Hospital, Byblos
  - Saint Joseph Hospital, Ed Daoura
  - Ain Wa Zein Hospital, El Chouf
  - Bellevue Medical Center, El- Metn
  - Hammoud Hospital, Saida
  - Haykal Hospital, Tripoli